CLINICAL TRIAL: NCT02558712
Title: Prospective Comparison of Technology-based Eye Care Services (TECS) With and Without OCT Assessment Versus Standard Face to Face Ophthalmologic Exam
Brief Title: Technology-based Eye Care Services (TECS) Compare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, April Maa, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00080630
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Cataract; Macular Degeneration; Glaucoma
Keywords: screening; tele-ophthalmology
MeSH Terms: conditions — Cataract; Macular Degeneration; Glaucoma | interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Face to face exam (Other): Standard of clinical care, 8 point eye exam
  Interventions: Other: Technology-based Eye Care Services (TECS) Protocol

INTERVENTIONS:
Other: Technology-based Eye Care Services (TECS) Protocol — Extensive History will be taken. Distance auto-refraction measurements will be made on both eyes. Eye pressure using the iCare tonometer and central corneal thickness (CCT) using the corneal pachymeter will be taken for each eye. Participants will have fundus photos taken following the standard VA diabetic teleretinal protocol. Then participants will have OCT Macula and Nerve performed. After protocol complete, then patients will see an ophthalmologist for standard eye exam.

SUMMARY:
The purpose of this study is to compare the Technology-based Eye Care Services (TECS) protocol to the standard face to face ophthalmologic exam.

DETAILED DESCRIPTION:
Patients will sign informed consent to enter the one visit study. They will undergo the study protocol and then see the face to face physician on the same day.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the Atlanta VA Medical Center (VAMC) New Comprehensive eye clinic

Exclusion Criteria:

* Known acute or chronic ocular issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2016-03; Primary Completion 2017-09 (Actual); Study Completion 2017-09-23 (Actual)

PRIMARY OUTCOMES:
Number of patients with accurate diagnosis of eye diseases from TECS protocol versus face to face eye exam with and without OCT | Evaluation Visit (Day 0)
  Clinical diagnosis in dichotomous (yes/no) decision tree. The clinical diagnosis of the TECS protocol readers will be compared to the face to face physician, with the face to face serving as the standard of care. The results will be done with and without OCT. Sensitivity, specificity, positive and negative predictive value will be calculated before and after OCT.

SECONDARY OUTCOMES:
Number of patients appropriately referred from the TECS protocol | Evaluation visit (Day 0)
  Total number of participants with a referral for face to face eye care with and without OCT
Number of participants with an accurate diagnosis for anterior segment disease | Evaluation visit (Day 0)
  The responses from an anterior segment questionnaire will be compared to the findings of the face to face physician exam for accuracy, using a (yes/no) decision tree. Sensitivity, specificity will be calculated using the face to face exam as the standard of care.
Inter-reader variability of the TECS protocol | Evaluation visit (Day 0)
  Kappa statistics reflecting the agreement between two readers on the same photo set of a single patient with and without OCT
Intra-reader variability of the TECS protocol | Evaluation visit (Day 0)
  Kappa statistics measuring agreement of the same reader reading the photographs of the same patient twice (after a washout period between photo reading sets) with and without OCT.

CONTACTS AND LOCATIONS:
Overall Officials: April Maa, MD, Principal Investigator — Emory University
Locations (1):
- Atlanta VA Medical Center, Decatur, Georgia, United States